CLINICAL TRIAL: NCT00903604
Title: Pharmacokinetics of AP214 Acetate in Patients Undergoing Cardiac Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Action Pharma A/S (Industry)
Responsible Party: Action Pharma A/S, Action Pharma A/S
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AP214-CS005
Record Dates: First submitted 2009-05-15; First posted 2009-05-18 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2011-05

CONDITIONS: Cardiac Surgery; Coronary Artery Bypass Grafting; Valve Surgery; Aortic Root or Ascending Aortic Aneurysm Repair Surgery
Keywords: Cardiac surgery; coronary artery bypass grafting; valve surgery; aortic root or ascending aortic aneurysm repair surgery; Acute kidney injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AP214 (Experimental): Infusions of sequential ascending dosages of AP214
  Interventions: Drug: AP214
- Placebo (Placebo Comparator): Infusions of saline solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AP214 — Three 10-minutes infusions of sequential ascending dosages of AP214
  Arms: AP214
Drug: Placebo — Three 10-minutes infusions of isotonic saline solution
  Arms: Placebo

SUMMARY:
The purpose of the present research study is to investigate the pharmacokinetics, as well as safety, tolerability and pharmacodynamics of different ascending dosing regimens of AP214 in patients undergoing cardiac surgery. AP214, the investigational drug, is being developed to potentially prevent post-surgical kidney injury after thoracic aortic aneurysm repair.

ELIGIBILITY:
Inclusion Criteria:

1. Has signed the trial-specific informed consent form.
2. Patients ≥ 18 years old, male or female, not of childbearing potential (postmenopausal or permanently sterilized, e.g. tubal ligation, hysterectomy, bilateral salpingectomy), regardless of ethnicity.
3. Patients undergoing CABG, valve(s), CABG/valve(s) and/or aortic root or ascending aortic aneurysm repair surgery.
4. Cleveland Clinic Renal Score ≥ 2 (higher than average risk for AKI).
5. EF ≥ 30%, evaluated within 2 months prior to screening visit.

Exclusion Criteria:

1. Cardiac surgery to be performed "off pump" without cardiopulmonary bypass.
2. Circulatory arrest in connection with aortic root or ascending aortic aneurysm repair surgery.
3. Confirmed or suspected endocarditis.
4. Requiring a reoperation on one of the valves within 3 months following the original valve surgical procedure.
5. Receiving Aprotinin during the trial, from Screening to Day 90.
6. Having undergone cardiovascular catheterization ≤ 48 hours prior to scheduled surgery.
7. Active peptic ulcer disease and gastritis.
8. Hemoccult positive stools, hematological, bleeding, and coagulation disorders.
9. Receiving dopamine at renal doses (2-4 mcg/kg/min), from Screening to Day of surgery.
10. S-Creatinine greater than 2.1 mg/dl.
11. Known or suspected hypersensitivity to the investigational medicinal product.
12. Known or suspected hypersensitivity to Ondansetron or other selective 5-hydroxytryptamine 3 (5-HT3) receptor antagonists.
13. Current participation in any other interventional clinical trial.
14. Previously dosed with AP214.
15. Use of investigational medicinal products within the previous 6 months.
16. Body weight above 140 kg.
17. History of any organ transplant.
18. Women who are of childbearing potential, pregnant, or breast-feeding.
19. Current abuse of alcohol or substance, according to the investigator's medical judgment.
20. Has a mental incapacity or language barriers precluding adequate understanding of trial procedures.
21. Is considered by the Investigator unsuitable to participate in the trial for any other reason, for instance due to a significant serious underlying condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2009-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To assess in patients the pharmacokinetics of AP214 administered as three 10-minute infusions in patients undergoing cardiac surgery. | Day 0 to Day 1
To assess the safety and tolerability of AP214, defined as a descriptive analysis of AEs and SAEs (including analysis of severity and relationship to trial drug) | Day 0-90

SECONDARY OUTCOMES:
To assess effect of AP214 on cardiac surgery induced systemic inflammation o determined by the post-operative peak plasma concentrations of TNF-α, IL-6, IL-8, and IL-10, and area under the curve (AUC) for TNF-α, IL-6, IL-8, and IL-10 | 0-24 hours
To assess effect of AP214 on development of post-surgical acute kidney injury (AKI), where AKI is evaluated by evaluation of serum creatinine values, urine output and renal replacement therapy free days. | Day 0 - Day 30
To assess the safety and tolerability of AP214 on standard safety laboratory data | Day 0-14
To assess the safety and tolerability of AP214 on vital signs | Day 0-90
To assess safety and tolerability of AP214 in terms of mortality by evaluation of overall mortality | Day 0-90
To assess the effect of AP214 at an organ level (CNS, heart, lung, and wound healing)as well as systemically. | Day 0-90

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Steinbrüchel, Professor, Principal Investigator — Department of Cardiac and Thoracic Surgery, Copenhagen University Hospital, Rigshospitalet
Locations (2):
- Denmark (2):
  - Department of Cardiac and Thoracic Surgery, Copenhagen University Hospital, Rigshospitalet, Copenhagen
  - Odense University Hospital, Department of Cardiac, Thoracic and Vascular Surgery, Odense